CLINICAL TRIAL: NCT06382701
Title: The Effect of Local Aromatherapy Applied to Hemodialysis Patients Before Arterio-venous Fistula Cannulation on Pain, Anxiety and Satisfaction
Brief Title: Effect of Aromatherapy on Pain, Anxiety and Satisfaction in Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Serife Cetin, doctor's degree, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Kayseri
Record Dates: First submitted 2024-04-17; First posted 2024-04-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hemodialysis Patients
Keywords: clove oil; arteriovenous fistula; pain; anxiety; satisfaction; hemodialysis
MeSH Terms: conditions — Arteriovenous Fistula; Pain; Anxiety Disorders; Personal Satisfaction | interventions — Aromatherapy

STUDY DESIGN:
Intervention Model Description: The study was designed as a randomized controlled and double-blind study to evaluate the effect of clove oil applied to arterio-venous fistula on pain and anxiety caused by cannulation and to determine the effect of the application on satisfaction.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Pre-cannulation spray application to the intervention and placebo groups will be provided by an interviewer trained by the researchers. Cannulations will be performed by nurses in the institution where the study is conducted. Data will be collected by the responsible nurses in the institutions.
  Patients participating in the study, researchers, and the nurse in charge will not know who is in the intervention and placebo groups.
  The research will be completed in twelve sessions over four weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): This is the group in which 0.5-1 ml of clove oil is applied as a spray to the arterio-venous fistula area, depending on the length of the fistula, ten minutes before needle cannulation in all hemodialysis sessions for four weeks in individuals receiving standard hemodialysis treatment.
  Interventions: Other: aromatherapy
- Placebo (Placebo Comparator): This is the group in which 0.5-1 ml of aromatic clove, which does not contain active ingredients and is dissolved in pure water, is applied as a spray to the arterio-venous fistula area, depending on the length of the fistula, ten minutes before needle cannulation in all hemodialysis sessions for four weeks in individuals receiving standard hemodialysis treatment.
  Interventions: Other: placebo

INTERVENTIONS:
Other: aromatherapy — Patients in the intervention group; ten minutes before the needle is inserted into the arterio-venous fistula, clove oil will be applied by the interviewer as a spray between 0.5-1 ml, depending on the length of the patient's fistula. Patients in the placebo group; 10 minutes before the needle is inserted into the arterio-venous fistula, 0.5-1 ml of aromatic cloves, which do not contain active ingredients and dissolved in pure water, will be applied as a spray by the interviewer, depending on the length of the patient's fistula.
  Arms: Intervention
Other: placebo — This is the group in which 0.5-1 ml of aromatic clove, which does not contain active ingredients and is dissolved in pure water, is applied as a spray to the arterio-venous fistula area, depending on the length of the fistula, ten minutes before needle cannulation in all hemodialysis sessions for four weeks in individuals receiving standard hemodialysis treatment.
  Arms: Placebo

SUMMARY:
The most active members of the healthcare professionals responsible for hemodialysis units are nurses, and they have a key role in pain, anxiety and satisfaction management as they are responsible for cannulation. Therefore, complementary and integrated practices need to be implemented based on evidence to strengthen the independent role of nurses in managing pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 18 years of age,
* Able to answer questions and communicate,
* No hearing, vision or speech impairments,
* Regularly undergoing hemodialysis three times a week,
* Having arterio-venous fistula for at least 3 months,
* Having pain during needle cannulation and scoring at least two or more points on the Visual Analogue Scale (VAS),
* Having been on hemodialysis for at least three months,
* Agreeing to participate in the study with their own consent,
* Patients who are not allergic to clove oil will be included in the study.

Exclusion Criteria:

* Having neuropathic pain,
* Patients with arterio-venous fistula and loss of sensation of more than 50% in the extremity,
* Patients with infection in the arterio-venous fistula line,
* Patients with aneurysm or pseudoaneurysm in arterio-venous fistula,
* Patients who have used analgesic medication/s in the last 6 hours,
* Patients who have used sedative agent(s) in the last 6 hours,
* Patients who used local anesthetic agents before needle intervention will not be included in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | before and after the intervention, for 1 month, 12 times
  This scale will be used in our study to evaluate the anxiety experienced by patients before needle cannulation and the pain and satisfaction experienced after needle cannulation.

SECONDARY OUTCOMES:
State and Trait Anxiety Inventory (STAI) | before and after the study, for 1 month, 2 times
  In our study, this scale will be used to evaluate the anxiety that patients may experience due to cannulation.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No